CLINICAL TRIAL: NCT05572567
Title: An Observational Study Within the CorEvitas Registry to Evaluate Safety and Effectiveness of Tofacitinib and Biologic Disease Modifying Antirheumatic Drugs (bDMARDs) in Japan Among Patients Treated for Moderately to Severely Active Rheumatoid Arthritis
Brief Title: Study to Evaluate Safety and Effects of Tofacitinib and Biologic Disease Modifying Antirheumatic Drugs in People Treated for Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921429
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Rheumatoid Arthritis (RA) patients treated with biologic and nonbiologic DMARDs: to include all Japanese patients taking Tofacitinib

SUMMARY:
This is a secondary structured database observational study conducted in Rheumatoid Arthritis (RA) patients treated with biologic and nonbiologic DMARDs, including tofacitinib, collected as part of the CorEvitas Japan RA Registry.

The data as of September 2022 will be used for this study. The study will include data from March 2016 to the latest data cut available in 2022 for both effectiveness and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Rheumatoid Arthritis (RA) according to the 1987 American College of Rheumatology (ACR) or the ACR/European Lead Against Rheumatism (EULAR) 2010 RA Classification Criteria;
* At least 18 years of age or older;
* Was / Must be prescribed or switching to the following eligible medication for the first time ever at the enrollment visit:
* csDMARD: methotrexate (closed in February 2018);
* Anti-TNF bDMARD: adalimumab (originator or biosimilar), certolizumab pegol, etanercept (originator or biosimilar), golimumab, infliximab (originator or biosimilar), or any other anti-TNF biosimilar approved during the study;
* Non-TNF bDMARD: abatacept, tocilizumab, sarilumab (closed in June 2020);
* JAK inhibitor: tofacitinib, baricitinib, peficitinib, filgotinib, upadacitinib.

Exclusion Criteria:

* Data that are prior to March 2016 and after June 2022

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in an existing registry database
Sampling Method: Non-Probability Sample
Enrollment: 1972 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Tanaka Y, Kishimoto M, Sonomoto K, Amano K, Harigai M, Onofrei A, O'Brien J, Margolin Z, Barr C, Mizuno Y, Agarwal E, Sugiyama N, Yamanaka H. Methotrexate, Tofacitinib, and Biologic Disease-Modifying Antirheumatic Drug Safety and Effectiveness Among Patients with Rheumatoid Arthritis in Japan: CorEvitas Registry Observational Study. Rheumatol Ther. 2024 Oct;11(5):1237-1253. doi: 10.1007/s40744-024-00700-2. Epub 2024 Jul 27. PMID 39066962
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective study of participants diagnosed with rheumatoid arthritis (RA) treated with biologic and nonbiologic disease-modifying antirheumatic drugs (DMARDs). Data was extracted from the CorEvitas Japan RA Registry from 01-Mar-2016 to 30-Jun-2022.
Groups:
- Methotrexate: Data of participants who had moderate to severe RA and treated with methotrexate was collected as part of CorEvitas Japan RA Registry from 01 March-2016 to 30-Jun-2022 and observed in this study.
- Tumor Necrosis Factor Inhibitors (TNFi): Data of participants who had moderate to severe RA and treated with TNFi was collected as part of CorEvitas Japan RA Registry from 01 March-2016 to 30-Jun-2022 and observed in this study.
- Non-TNFi: Data of participants who had moderate to severe RA and treated with non-TNFi was collected as part of CorEvitas Japan RA Registry from 01 March-2016 to 30-Jun-2022 and observed in this study.
- Tofacitinib: Data of participants who had moderate to severe RA and treated with tofacitinib was collected as part of CorEvitas Japan RA Registry from 01 March-2016 to 30-Jun-2022 and observed in this study.
Period: Overall Study
Arm/Group | Methotrexate | Tumor Necrosis Factor Inhibitors (TNFi) | Non-TNFi | Tofacitinib
Started | 298 | 663 | 758 | 253
Completed | 298 | 663 | 758 | 253
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Tumor Necrosis Factor Inhibitors (TNFi) | Non-TNFi | Tofacitinib | Total
Number analyzed (Participants) | 298 | 663 | 758 | 253 | 1972
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (14.0) | 60.3 (15.1) | 65.8 (12.6) | 62.1 (13.2) | 62.6 (14.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 222 | 538 | 582 | 208 | 1550
  Male | 76 | 125 | 176 | 45 | 422
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 295 | 655 | 750 | 249 | 1949
  Unknown or not reported | 3 | 8 | 8 | 4 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Incidence Rate of Total Cardiovascular Disease (CVD) Events
Description: Incidence rate was defined as participants with total CVD events per (/) 100 person years. Total CVD was defined as hypertension requiring hospitalization, cardiac revascularization procedure (CABG, stent, angioplasty), ventricular arrhythmia, cardiac arrest, myocardial infarction, acute coronary syndrome, unstable angina, congestive heart failure (CHF) requiring hospitalization, stroke, transient ischemic attack, other cardiovascular event (specify), deep vein thrombosis, peripheral arterial thromboembolic event, urgent peripheral arterial revascularization, peripheral ischemia or gangrene (necrosis) and pulmonary embolism. Index visit was defined as the initiation date of the therapy of interest. Mean of incidence rate of total CVD events was calculated and reported.
Time Frame: Retrospective data collection from index visit date up to follow-up or latest data cut on 30 June 2022 (Approximately up to 75 months)
Population: Participants who had RA and initiated treatment with methotrexate, tofacitinib, TNFi or non-TNFi and who were followed up after first dose of the drug were included. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Participants with event/100 Person years
Groups:
- TNFi: Data of participants who had moderate to severe RA and treated with TNFi was collected as part of CorEvitas Japan RA Registry from 01 March-2016 to 30-Jun-2022 and observed in this study.
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 4 | 11 | 23 | 8
Participants with event/100 Person years | 0.51 [0.01 to 1] | 0.76 [0.31 to 1.21] | 1.4 [0.83 to 1.97] | 1.54 [0.47 to 2.61]

2. Primary Outcome: Mean Incidence Rate of Serious Infections Events
Description: Incidence rate was defined as mean number of participants with serious infection events per 100 person years. Total serious infections were defined as infections meeting serious adverse event criteria or which required treatment with intravenous (IV) antibiotics. Serious infection types collected in the registry were pneumonia, sepsis, joint/bursa, cellulitis/skin, sinusitis, diverticulitis, bronchitis, gastroenteritis, meningitis/encephalitis, urinary tract infection, upper respiratory infection, active tuberculosis and other serious infections. Mean of incidence rate of total serious infection events was calculated and reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Participants with event/100 Person years
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 15 | 37 | 79 | 16
Participants with event/100 Person years | 1.94 [0.96 to 2.92] | 2.61 [1.77 to 3.45] | 5.02 [3.91 to 6.12] | 3.1 [1.58 to 4.61]

3. Primary Outcome: Mean Incidence Rate of Total Herpes Zoster Events
Description: Incidence rate was defined as mean number of participants with total Herpes Zoster events per 100 person years. Total herpes zoster included both serious and non-serious herpes zoster events. Mean of incidence rate of total herpes zoster events was calculated and reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Participants with event/100 Person years
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 7 | 20 | 35 | 39
Participants with event/100 Person years | 0.9 [0.23 to 1.57] | 1.39 [0.78 to 2] | 2.18 [1.46 to 2.9] | 8.07 [5.53 to 10.58]

4. Primary Outcome: Mean Incidence Rate of Total Malignancy Excluding Non-Melanoma Skin Cancer (NMSC)
Description: Incidence rate (number of participants with event per 100 person year) was defined as the mean number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. Total malignancy excluding non-melanoma skin cancer included lymphoma, lung cancer, breast cancer, skin cancer (melanoma), and other cancers. Mean of incidence rate of total malignancy excluding non-melanoma skin cancer was calculated and reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Participants with event/100 Person years
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 19 | 33 | 41 | 11
Participants with event/100 Person years | 1.72 [0.95 to 2.5] | 1.71 [1.13 to 2.29] | 1.93 [1.34 to 2.51] | 1.51 [0.62 to 2.41]

5. Primary Outcome: Mean Change From Baseline in Clinical Disease Activity Index (CDAI) at 6 Months
Description: CDAI was the numerical sum of four outcome parameters: Tender joint count (TJC) or swollen joint count (SJC) both based on a 28-joint assessment, participant's assessment (PtGA) of disease activity and physician's global assessment (PGA) of disease activity both assessed on a 0 to 10 centimeter (cm) visual analogue scale (VAS) (higher scores indicated greater affection due to disease activity). CDAI total score ranged from 0 to 76. Higher scores indicated greater affection due to disease activity. CDAI less than or equal to (<=) 2.8 indicated disease remission, greater than (>) 2.8 to 10 indicated low disease activity, >10 to 22 indicates moderate disease activity, and >22 indicated high disease activity. Mean change from baseline was calculated by subtracting the baseline value from the 6-month value.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: Participants who had RA and initiated treatment with methotrexate, tofacitinib, TNFi or non-TNFi and who were followed up after first dose of the drug were included.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Units on a scale | -10.1 [-11.5 to -8.5] | -10.4 [-11.5 to -9.4] | -11.5 [-12.5 to -10.6] | -11.7 [-13.4 to -9.9]

6. Primary Outcome: Mean Change From Baseline in Japanese Health Assessment Questionnaire (J-HAQ) at 6 Months
Description: HAQ: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom, arise, eat, walk, reach, grip, hygiene, and common activities over past week. Each item scored on 4-point scale, 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3: 0=least difficulty and 3=extreme difficulty. Higher scores indicated worse functioning. Mean change from baseline was calculated by subtracting the baseline value from the 6-month value.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Units on a scale | -0.3 [-0.4 to -0.2] | -0.2 [-0.3 to -0.2] | -0.3 [-0.3 to -0.2] | -0.3 [-0.4 to -0.2]

7. Primary Outcome: Mean Change From Baseline in Participant's Pain at 6 Months
Description: Participants were asked the following question to answer on a numeric rating scale (NRS): "How much pain have you had because of your arthritis in the past week?" The scale ranged from 0-100, where 0=no pain and 100=pain as bad as it could be. Higher scores indicated worsening of condition. Mean change from baseline in participant's pain was calculated and reported.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Units on a scale | -21.7 [-25.1 to -18.3] | -17.6 [-19.9 to -15.3] | -17.4 [-19.5 to -15.2] | -21.4 [-25.4 to -17.5]

8. Primary Outcome: Mean Change From Baseline in Participant's Fatigue at 6 Months
Description: Visual Analogue Scale (VAS) was a standardized tool for measuring overall health. Participants recorded their fatigue score on a range of 0 to 100, where higher score indicated higher intensity of fatigue. Mean change from baseline in participant's fatigue was calculated and reported.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Units on a scale | -13 [-16.3 to -9.9] | -9.4 [-11.6 to -7.2] | -10.7 [-12.8 to -8.7] | -15.5 [-19.2 to -11.8]

9. Primary Outcome: Mean Change From Baseline in Participant's Global Assessment at 6 Months
Description: Participant's global assessment of disease activity on a 100 millimeter (mm) Visual Analog Scale (VAS) (scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicated worse health condition). Mean change from baseline was calculated by subtracting the baseline value from the 6-month value.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
mm | -18.5 [-21.8 to -15.2] | -16.8 [-19.1 to -14.6] | -16.1 [-18.2 to -14.0] | -19.5 [-23.4 to -15.7]

10. Primary Outcome: Mean Change From Baseline in Morning Stiffness at 6 Months
Description: CDAI and other continuous measures like morning stiffness were represented as mean change from baseline to 6-months and were calculated by subtracting the baseline value from the 6-month value.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Minutes | -31.5 [-35.9 to -27.1] | -22.4 [-25.4 to -19.5] | -17.9 [-20.6 to -15.1] | -19.7 [-24.7 to -14.6]

11. Primary Outcome: Change in Percentage of Participants Reporting Moderate/Severe/Extreme Difficulty Levels for EQ-5D-5L From Baseline at Month 6
Description: EQ-5D-5L was a participant rated questionnaire to assess health-related quality of life. It assessed level of current health in 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each domain had 5 levels: 1= no problems, 2=slight problems, 3=moderate problems, 4=severe problems, or 5=extreme problems/unable to do task. Total score for each domain was from 1-5, where higher levels/scores indicated more difficulty in each domain. At baseline and 6 months, percentage of participants who recorded "moderate", "severe" or "extreme problems" level in each of the domain were assessed; then change was calculated in percentage of participants from baseline at Month 6 and was reported in this outcome measure.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Percentage of participants
  Mobility | -10.2 [-14.0 to -6.5] | -6.8 [-9.4 to -4.3] | -11.1 [-13.4 to -8.7] | -10.8 [-15.2 to -6.4]
  Selfcare | -8.6 [-12.0 to -5.2] | -7.6 [-9.9 to -5.3] | -12.2 [-14.3 to -10.0] | -9 [-12.9 to -5.0]
  Usual activities | -12.6 [-16.5 to -8.7] | -13.5 [-16.2 to -10.8] | -14.5 [-17.0 to -12.0] | -14.8 [-19.3 to -10.3]
  Pain/discomfort | -31.2 [-35.9 to -26.4] | -24.6 [-27.9 to -21.4] | -28.5 [-31.5 to -25.5] | -25.3 [-30.8 to -19.8]
  Depression/anxiety | -9.5 [-12.9 to -6.0] | -7.1 [-9.5 to -4.7] | -9.5 [-11.7 to -7.3] | -4.2 [-8.2 to -0.2]

12. Primary Outcome: Percentage of Participants Who Achieved Minimally Clinically Important Difference (MCID) Improvement at 6 Months
Description: MCID improvement assessed based on CDAI. CDAI: numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; CDAI total score = 0-76, higher scores=greater affection due to disease activity (DA). CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low DA, >10 to 22 = moderate DA, and >22 = high DA. MCID improvement defined by difference in CDAI from baseline (at time of tofacitinib initiation) to 6-month visit.
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Percentage of Participants | 61.1 [55.3 to 66.9] | 57.6 [53.6 to 61.7] | 65 [61.3 to 68.6] | 65.1 [58.4 to 71.8]

13. Primary Outcome: Percentage of Participants Who Achieved Modified American College of Rheumatology (mACR) 20 Response Score at 6 Months
Description: mACR20 response: >= 20 percent (%) improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the j-HAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: The participants who had RA and initiated treatment with methotrexate, tofacitinib, TNFi or non-TNFi and who were followed up after first dose of the drug were included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Percentage of Participants | 47.1 [41.2 to 53.0] | 39.8 [35.9 to 43.7] | 45.6 [41.8 to 49.3] | 44.4 [37.6 to 51.2]

14. Primary Outcome: Percentage of Participants Who Achieved mACR 50 Response Score at 6 Months
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the j-HAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Percentage of Participants | 35.9 [30.2 to 41.5] | 29.9 [26.2 to 33.5] | 31.7 [28.3 to 35.2] | 33.2 [26.7 to 39.6]

15. Primary Outcome: Percentage of Participants Who Achieved mACR 70 Response Score at 6 Months
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the j-HAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: Baseline, Month 6 (Retrospective data collection from 01 March-2016 to 30-Jun-2022)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Methotrexate | TNFi | Non-TNFi | Tofacitinib
Number analyzed (Participants) | 276 | 603 | 687 | 205
Percentage of Participants | 21.4 [16.5 to 26.2] | 18.2 [15.2 to 21.3] | 18.6 [15.7 to 21.5] | 22.4 [16.7 to 28.1]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From date of RA diagnosis until the end of follow-up (approximately up to 75 months, retrospective data collection from 01 March-2016 to 30-Jun-2022). Data for non-serious adverse events (SAEs) and SAEs were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs.
Description: This study involves data that exist as structured data by the time of study start. In these data sources, it was not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable participant, identifiable reporter, a suspect product, and event) cannot be met.
Arm/Group | Methotrexate | Tumor Necrosis Factor Inhibitors (TNFi) | Non-TNFi | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/663 | 0/758 | 0/253
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT05572567/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT05572567/SAP_001.pdf